CLINICAL TRIAL: NCT05469412
Title: To Compare Pharmacological and Non-Pharmacological Interventions (Use of Technology) For Alleviating Preoperative Anxiety In Children Undergoing General Anesthesia In A Tertiary Care Hospital Of Pakistan: A Randomized Controlled Trial.
Brief Title: Comparison of Pharmacological and Non-Pharmacological Interventions For Alleviating Preoperative Anxiety In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Asghar Ali, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-7684-21894
Record Dates: First submitted 2022-06-13; First posted 2022-07-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Anxiety and Fear
Keywords: Preoperative Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Vaginal Creams, Foams, and Jellies; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Standard management combined with distraction by using technology (Tablets/iPads).
  Interventions: Device: iPad®
- Control group (Active Comparator): Standard management combined with pharmacological intervention (oral midazolam 0.5 mg/kg) administered at least 30 min before surgery (maximum 20mg).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Device: iPad® — Use of Technology.
  Other Names: Tablet
  Arms: Interventional group
Drug: Midazolam — Standard management combined with pharmacological intervention (oral midazolam 0.5 mg/kg) administered at least 30 min before surgery (maximum 20mg).
  Arms: Control group

SUMMARY:
The purpose of this study is to find out any beneficial effects of electronic devices over preoperative pharmacological intervention in the preoperative period.

DETAILED DESCRIPTION:
Preparation for surgery with the induction of general anesthesia can be a stressful experience for a child. Preoperative anxiety can prolong induction of anesthesia and postoperative recovery, as well as increasing the risk of postoperative delirium, pain, and analgesic use.

Pharmacological interventions are associated with increased cost to the hospital, potential surgical delay while waiting for the medication to take effect, and delayed discharge from the recovery room. Non-pharmacological modalities comprise education, behavioral techniques, parental presence at induction of anesthesia, and using technology including cellular phones and tablets/iPad, with each category including an array of effective strategies for reducing anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 2 and 12 years old
2. ASA I and II
3. Informed consent signed by parents or legal guardians

Exclusion Criteria:

1. Previous exposure to surgery
2. Contraindication to midazolam
3. Patients with developmental delay
4. Patients with significant visual/hearing problems

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale | Day 1
  The instrument contains 27 items in 5 categories that indicate preoperative anxiety in children: activity, emotional expressivity, state of arousal, vocalization, and use of parents.
  Scores range from 23.33 to 100, with higher values indicating higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manyande A, Cyna AM, Yip P, Chooi C, Middleton P. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD006447. doi: 10.1002/14651858.CD006447.pub3. PMID 26171895
- [Background] Agbayani CG, Fortier MA, Kain ZN. Non-pharmacological methods of reducing perioperative anxiety in children. BJA Educ. 2020 Dec;20(12):424-430. doi: 10.1016/j.bjae.2020.08.003. Epub 2020 Oct 21. No abstract available. PMID 33456927
- [Background] Cheng X, Chen Z, Zhang L, Xu P, Qin F, Jiao X, Wang Y, Lin M, Zeng L, Huang L, Yu D. Efficacy and Safety of Midazolam Oral Solution for Sedative Hypnosis and Anti-anxiety in Children: A Systematic Review and Meta-Analysis. Front Pharmacol. 2020 Mar 18;11:225. doi: 10.3389/fphar.2020.00225. eCollection 2020. PMID 32256348